CLINICAL TRIAL: NCT04209335
Title: Isometric Core Muscle Endurance in Healthy Active and Non-active Working Age Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanna Holmberg (Other)
Collaborators: University of Salford (Other)
Responsible Party: Sponsor-Investigator, Hanna Holmberg, student of MSc, University of Salford
Organization: University of Salford (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HST 1718-316
Record Dates: First submitted 2019-12-16; First posted 2019-12-24 (Actual); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Physical Endurance
Keywords: aging; lower back pain; physical activity level; body mass index; core muscle endurance; gender; McGill V-sit; Biering-Sorensen; sideplank
MeSH Terms: conditions — Low Back Pain; Coitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy working age population (Other): isometric core muscle endurance tests (McGill V-sit, Biering-Sorensen and sideplank)
  Interventions: Other: isometric core muscle endurance testing

INTERVENTIONS:
Other: isometric core muscle endurance testing — holding previously described isometric positions until fatigue

SUMMARY:
Objectives: The purpose of this study was to investigate a possible correlation between core muscle endurance and participants' age in healthy adult population. Secondary purpose was to identify other dependent variables influencing isometric core muscle endurance (e.g. low back pain, physical activity, gender, body mass index).

Methods: 48 (35 females, 13 males) healthy adults (aged 21-66 years) performed 4 isometric core muscle endurance tests- Biering-Sorensen, McGill V-sit, right and left side plank. A correlation between core endurance and age, gender, lower back pain (LBP), physical activity level (PAL), and body mass index (BMI) was calculated.

DETAILED DESCRIPTION:
This is the first study to investigate the core muscle endurance of different age groups and genders with all four endurance tests of the core.

Since strength and endurance are key to keeping healthy as we age and National Institute for Health and Care Excellence (NICE) and European guidelines advocate them, this study aims to look at the 3 main measurements of core endurance namely flexor, extensor and lateral muscles, and the possible correlations with age, PAL, existence of LBP, BMI and gender. Each participant performed 4 isometric core endurance tests in the same order- 1. Biering-Sorensen, 2.-3. side plank on both sides, and 4. McGill V-sit. All participants were tested by the same tester to reduce potential differences in procedure and testing error. The four tests were each measured using a stopwatch and documented in seconds. Each participant was told the time they had reached during testing to improve their motivation. Pain during testing was documented.

Based on the normative data of abdominal muscle endurance for young adults Null hypothesis (H0)- There is no significant difference in endurance tests for age, presence of LBP or PAL. Hypothesis (H1)- Any significant difference in endurance tests for age, presence of LBP or PAL are due to chance factors. This is a two-tailed hypothesis, as previous evidence shows conflicting results. Pearson's correlation and Independent T-test in SPSS (The Statistical Package for the Social Sciences) were used to confirm or reject the possible correlations between the core muscle endurance and age, LBP, PAL, gender, BMI, and participants' job.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-70 (working age population)
* healthy
* active and non-active
* with or without non-specific lower back pain

Exclusion Criteria:

* all serious pathologies and diagnosis that could affect the ability to perform the tests safely including acute pain, neurological, musculoskeletal, cardiovascular diseases, spinal pathologies (e.g. spondylitis, acute herniated disc, cauda equina, hypertension, epilepsy, tumour, previous fracture or surgery in trunk, structured deformity, osteoporosis)
* sudden change in health
* personal reasons
* severe pain during testing
* competing in any sports higher than amateur level

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynne E Gaskell, MSc, Principal Investigator — Supervisor; Hanna Holmberg, MSc, Principal Investigator — student
Locations (1):
- University of Salford, Manchester, Salford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the general population with different lifestyles and jobs.
Period: Overall Study
Arm/Group | Healthy Working Age Population
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Healthy Working Age Population
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants] — Participants were viewed separately as well as in two groups- participants up to 40 years and participants over 40 years.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 47
    >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 40 [21 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Inter-Quartile Range); unit: Kg/m^2] | 23.8 [15.9 to 31.6]
Number of participants considered active [Count of Participants; unit: Participants] — Based on national and international guidelines. It is suggested that adults aged between 18 and 65 should do moderate-intensity aerobic physical activities for a minimum of 30 minutes, 5 times a week, or high-intensity aerobic activities 20 minutes, 3 times a week. Participants who met the above guideline were considered as active.
  Participants | 27
Number of participants who have experienced non-specific lower back pain [Count of Participants; unit: Participants] — Participants were asked if they have experienced non-specific lower back pain in last 6 months.
  Participants | 15

OUTCOME MEASURES:

1. Primary Outcome: Core Muscle Endurance
Description: time in seconds after summing the results of all 4 tests
Time Frame: at the time of testing, in 1 hour
Measure: Mean (Standard Error); unit: seconds
Groups:
- Healthy Working Age Population: the sum of 4 isometric core muscle endurance tests (McGill V-sit, Biering-Sorensen and sideplank on each side)
  isometric core muscle endurance testing: holding previously described isometric positions until fatigue
Arm/Group | Healthy Working Age Population
Number analyzed (Participants) | 48
seconds | 530.5 (34.6)

2. Secondary Outcome: Body Mass Index
Description: weight(kg)/height(cm)2 Value under 18.5 is considered underweight, over 25 overweight, and over 30 obese.
Time Frame: during the time of testing, in 1 h
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Groups:
- Healthy Working Age Population: the body mass index of the participant, at the time of testing
Arm/Group | Healthy Working Age Population
Number analyzed (Participants) | 48
units on a scale | 23.8 [15.9 to 31.6]

3. Secondary Outcome: Physical Activity Level Questionnaire
Description: physical activity level based on national and international recommendations
Time Frame: at the time of testing, last 2 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Healthy Working Age Population: Number of active participants who met national and international guidelines
Arm/Group | Healthy Working Age Population
Number analyzed (Participants) | 48
Participants | 27

4. Secondary Outcome: Number of Participants Who Have Experienced Non-specific Lower Back Pain
Description: categorical data, experience of nonspecific low back pain up to 6 months before the assessment
Time Frame: up to 6 months before the assessment
Measure: Count of Participants; unit: Participants
Groups:
- Healthy Working Age Population: Number of participants who have experienced nonspecific low back pain
Arm/Group | Healthy Working Age Population
Number analyzed (Participants) | 48
Participants | 15

ADVERSE EVENTS:
Time Frame: Data was collected on a nonspecific time of the day, in 1 hour
Description: All possible health risks were excluded in recruitment phase as it was considered as exclusion criteria. Also, each participant was allowed to stop at any time during the testing. All possible other events were recorded from participants' feedback during and right after testing.
Arm/Group | Healthy Working Age Population
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 12/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Working Age Population (N=48)
Shoulder, elbow, lower back pain (Musculoskeletal and connective tissue disorders) | 12 (12) — Pain during testing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT04209335/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT04209335/ICF_001.pdf